CLINICAL TRIAL: NCT02705755
Title: A Phase 2 Study to Assess the Effect of TD-9855 in Subjects With Neurogenic Orthostatic Hypotension
Brief Title: TD-9855 Phase 2 in Neurogenic Orthostatic Hypotension (nOH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0145
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Results first posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-02

CONDITIONS: Neurogenic Orthostatic Hypotension; Multiple System Atrophy (MSA) With Orthostatic Hypotension; Pure Autonomic Failure; Parkinson Disease; Hypotension, Orthostatic; Orthostatic Hypotension; Pure Autonomic Failure With Orthostatic Hypotension; Parkinson Disease With Orthostatic Hypotension
Keywords: Neurogenic Orthostatic Hypotension (nOH); Multiple System Atrophy (MSA); Pure Autonomic Failure; Parkinson Disease(PD); nOH; MSA; PD; PAF; Orthostatic Hypotension; ampreloxetine; TD-9855
MeSH Terms: conditions — Multiple system atrophy (MSA) with orthostatic hypotension; Pure Autonomic Failure; Parkinson Disease; Hypotension, Orthostatic; Multiple System Atrophy | interventions — ampreloxetine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TD-9855 Part A (Experimental): Subjects will receive placebo and escalating single doses of TD-9855
  Interventions: Drug: TD-9855; Drug: Placebo
- TD-9855 Part B (Experimental): Subjects will receive a single dose of TD-9855 or placebo.
  Interventions: Drug: TD-9855; Drug: Placebo
- TD-9855 Part C (Experimental): Subjects will receive once daily doses of TD-9855 for up to 5 months as part of an optional outpatient open-label extension arm.
  Interventions: Drug: TD-9855; Drug: Placebo

INTERVENTIONS:
Drug: TD-9855 — Administered orally.
Drug: Placebo — Administered orally.

SUMMARY:
This multiple-center, 3-part, single-blind dose escalation (Part A), randomized, double-blind (Part B), and open-label multiple dose extension (Part C) study will be conducted in male and female subjects with neurogenic orthostatic hypotension to evaluate the effect of TD-9855 in improving symptoms of orthostatic intolerance.

DETAILED DESCRIPTION:
Part A followed a daily, single-escalating-dose design, starting with placebo on Day 1, followed by a dose of 2.5 mg TD-9855 on Day 2, and proceeding to higher daily doses of TD-9855 up to a maximum dose of 20 mg based on safety, tolerability, and determination of a pressor effect.

The starting dose in Part A was initially set to 1 mg (Day 2), escalating to a maximum dose of 10 mg (Day 5), but this was revised to start at 2.5 mg (Day 2) and escalate to 20 mg (Day 5) in protocol amendment 2 (Section 9.8.1).

Part B followed a randomized, placebo-controlled, parallel design, evaluating an acute dose of TD-9855 that was determined to have a pressor effect and to be generally well tolerated for a given subject from Part A.

Subjects who completed Part A, demonstrated a pressor effect in Part A, and remained otherwise eligible, had the option to receive open-label TD-9855 by tablet daily for up to 5 months (20 weeks) during Part C.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic orthostatic hypotension due to Parkinson's disease, multiple system atrophy, or pure autonomic failure, (i.e. neurogenic orthostatic hypotension).
* At screening, subject must meet the diagnostic criteria of neurogenic orthostatic hypotension, as demonstrated by a ≥ 30 mm Hg drop in systolic blood pressure (SBP) within 5 minutes of standing.
* Impaired autonomic reflexes, as determined by absence of BP overshoot during phase IV of the Valsalva maneuver, in subjects where Valsalva is performed, as appropriate.
* For the optional open-label extension study subjects must have demonstrated a pressor effect and completed dosing in Part A.

Exclusion Criteria:

* Systemic illnesses known to produce autonomic neuropathy, including but not limited to diabetes mellitus, amyloidosis, monoclonal gammopathy of unknown significance, and autoimmune neuropathies.
* Concomitant use of vasoconstricting agents for the purpose of increasing BP such as ephedrine, dihydroergotamine, or midodrine must be stopped at least 2 days or five half lives (whichever is longer) prior to dosing on Day 1 of Part A and C, and throughout the duration of Part C. Subjects previously enrolled in Part A under previous versions of the protocol will continue taking fludrocortisone during the washout period and in Part C at the dose and regimen used in Part A. For new subjects enrolling in Part A under Amendment 3, fludrocortisone use in both Parts of the study and during the washout period will be limited to 0.1 mg QD.
* Concomitant use of anti-hypertensive medication for the treatment of essential hypertension unrelated to autonomic dysfunction.
* Known or suspected alcohol or substance abuse within the past 12 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma, US, Inc.
Locations (6):
- United States (6):
  - Theravance Biopharma Investigational Site, Long Beach, California
  - Theravance Biopharma Investigational Site, Farmington Hills, Michigan
  - Theravance Biopharma Investigational Site, Berlin, New Jersey
  - Theravance Biopharma Investigational Site, New York, New York
  - Theravance Biopharma Investigational Site, Nashville, Tennessee
  - Theravance Biopharma Investigational Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaufmann H, Vickery R, Wang W, Kanodia J, Shibao CA, Norcliffe-Kaufmann L, Haumann B, Biaggioni I. Safety and efficacy of ampreloxetine in symptomatic neurogenic orthostatic hypotension: a phase 2 trial. Clin Auton Res. 2021 Dec;31(6):699-711. doi: 10.1007/s10286-021-00827-0. Epub 2021 Oct 17. PMID 34657222
- [Derived] Lo A, Norcliffe-Kaufmann L, Vickery R, Bourdet D, Kanodia J. Pharmacokinetics and pharmacodynamics of ampreloxetine, a novel, selective norepinephrine reuptake inhibitor, in symptomatic neurogenic orthostatic hypotension. Clin Auton Res. 2021 Jun;31(3):395-403. doi: 10.1007/s10286-021-00800-x. Epub 2021 Mar 29. PMID 33782836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 participants were enrolled across 6 sites in the United States between September 2017 and November 2018.
Pre-assignment Details: 34 participants were screened and all were enrolled and treated with study drug.
Groups:
- Part A: Dose Escalation (Within Group): Part A of this study was a single blind within group dose escalation design. It started with placebo on Day 1 followed by a dose of 2.5 mg TD-9855 on Day 2, and proceeded to higher daily doses of TD-9855 up to maximum dose of 20 mg on Day 5 depending on safety, tolerability, and determination of a pressor effect.
  There was a washout period of a minimum of 8 days up to 36 days between Part A and Part B and a minimum of 8 days between Part A and Part C.
- Part B: Randomized - Placebo: Part B of this study followed a randomized, double-blind, placebo-controlled, parallel design at the dose level of TD-9855 determined to have a pressor effect for a given participant in Part A. Participants from Part A were rolled over into Part B.
  Following the washout period after Part A, participants were randomized to receive a single dose of placebo on Day 1 of the treatment period.
- Part B: Randomized- TD-9855: Part B of this study followed a randomized, double-blind, placebo-controlled, parallel design at the dose level of TD-9855 determined to have a pressor effect for a given participant in Part A. Participants from Part A were rolled over into Part B.
  Following the washout period after Part A, participants were randomized to receive a single dose of their previously tolerated dose of TD-9855 on Day 1 of the treatment period.
- Part C: Dose Extension: Part C of this study was an open-label dose extension period. Participants who completed Part A, demonstrated a pressor effect in Part A, and remained otherwise eligible, had the option to receive open-label TD-9855 daily for up to 20 weeks in Part C.
  The dose of TD-9855 administered on Day 1 in Part C, following the washout period, was equal to 50% (or lower) of the highest tolerated dose administered during Part A. After Day 29, dose increases were made at the discretion of the investigator.
Period: Part A (6 Days)
Arm/Group | Part A: Dose Escalation (Within Group) | Part B: Randomized - Placebo | Part B: Randomized- TD-9855 | Part C: Dose Extension
Started (Each participant was titrated to their individual maximum tolerated dose.) | 34 | 0 | 0 | 0
Participants Who Received Placebo | 34 | 0 | 0 | 0
Participants Who Received 1 mg Study Drug (Participants who were enrolled prior to protocol amendment 2 received a starting dose of 1 mg TD-9855 as an oral solution on Day 2 of Part A and escalated to 10 mg. Beginning with protocol amendment 2, the starting dose was changed to 2.5 mg with dose escalation to 20 mg.) | 17 | 0 | 0 | 0
Participants Who Received 2.5 mg Study Drug | 31 | 0 | 0 | 0
Participants Who Received 5 mg Study Drug | 29 | 0 | 0 | 0
Participants Who Received 10 mg Study Drug | 28 | 0 | 0 | 0
Participants Who Received 20 mg Study Drug | 13 | 0 | 0 | 0
Participants Who Rolled to Part B | 10 | 0 | 0 | 0
Participants Who Rolled to Part C | 21 | 0 | 0 | 0
Completed | 29 | 0 | 0 | 0
Not Completed | 5 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Part B (1 Day)
Arm/Group | Part A: Dose Escalation (Within Group) | Part B: Randomized - Placebo | Part B: Randomized- TD-9855 | Part C: Dose Extension
Started | 0 | 5 | 5 (Each participant received their individual maximum tolerated dose from Part A.) | 0
Received Study Drug | 0 | 5 | 5 | 0
Completed | 0 | 5 | 5 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part C (20 Weeks)
Arm/Group | Part A: Dose Escalation (Within Group) | Part B: Randomized - Placebo | Part B: Randomized- TD-9855 | Part C: Dose Extension
Started | 0 | 0 | 0 | 21
Received Study Drug | 0 | 0 | 0 | 21
Completed | 0 | 0 | 0 | 11
Not Completed | 0 | 0 | 0 | 10
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants from Parts A, B, and C. Each part of the study is reported as a row in each of the Baseline Measures.
Arm/Group | All Study Participants
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number analyzed in each row is based on the number of participants enrolled in that part of the study.
  years
    Part A: Dose Escalation (Within Group) | 65.8 (7.94)
    Part B: Randomized - Placebo: number analyzed (Participants) | 5
    Part B: Randomized - Placebo | 65.2 (8.98)
    Part B: Randomized - TD-9855: number analyzed (Participants) | 5
    Part B: Randomized - TD-9855 | 66.4 (5.22)
    Part C: Dose Extension: number analyzed (Participants) | 21
    Part C: Dose Extension | 64.1 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analyzed in each row is based on the number of participants enrolled in that part of the study.
  Participants
    Part A: Part A: Dose Escalation (Within Group): Female | 12
    Part A: Part A: Dose Escalation (Within Group): Male | 22
    Part B: Randomized - Placebo: number analyzed (Participants) | 5
    Part B: Randomized - Placebo: Female | 2
    Part B: Randomized - Placebo: Male | 3
    Part B: Randomized - TD-9855: number analyzed (Participants) | 5
    Part B: Randomized - TD-9855: Female | 2
    Part B: Randomized - TD-9855: Male | 3
    Part C: Dose Extension: number analyzed (Participants) | 21
    Part C: Dose Extension: Female | 9
    Part C: Dose Extension: Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: The number analyzed in each row is based on the number of participants enrolled in that part of the study.
  Participants
    Part A: Dose Escalation (Within Group): Hispanic or Latino | 3
    Part A: Dose Escalation (Within Group): Not Hispanic or Latino | 30
    Part A: Dose Escalation (Within Group): Unknown or Not Reported | 1
    Part B: Randomized - Placebo: number analyzed (Participants) | 5
    Part B: Randomized - Placebo: Hispanic or Latino | 1
    Part B: Randomized - Placebo: Not Hispanic or Latino | 4
    Part B: Randomized - Placebo: Unknown or Not Reported | 0
    Part B: Randomized - TD-9855: number analyzed (Participants) | 5
    Part B: Randomized - TD-9855: Hispanic or Latino | 0
    Part B: Randomized - TD-9855: Not Hispanic or Latino | 5
    Part B: Randomized - TD-9855: Unknown or Not Reported | 0
    Part C: Dose Extension: number analyzed (Participants) | 21
    Part C: Dose Extension: Hispanic or Latino | 2
    Part C: Dose Extension: Not Hispanic or Latino | 18
    Part C: Dose Extension: Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: The number analyzed in each row is based on the number of participants enrolled in that part of the study.
  Participants
    Part A: Dose Escalation (Within Group): American Indian or Alaska Native | 0
    Part A: Dose Escalation (Within Group): Asian | 1
    Part A: Dose Escalation (Within Group): Native Hawaiian or Other Pacific Islander | 0
    Part A: Dose Escalation (Within Group): Black or African American | 2
    Part A: Dose Escalation (Within Group): White | 31
    Part A: Dose Escalation (Within Group): More than one race | 0
    Part A: Dose Escalation (Within Group): Unknown or Not Reported | 0
    Part B: Randomized - Placebo: number analyzed (Participants) | 5
    Part B: Randomized - Placebo: American Indian or Alaska Native | 0
    Part B: Randomized - Placebo: Asian | 1
    Part B: Randomized - Placebo: Native Hawaiian or Other Pacific Islander | 0
    Part B: Randomized - Placebo: Black or African American | 0
    Part B: Randomized - Placebo: White | 4
    Part B: Randomized - Placebo: More than one race | 0
    Part B: Randomized - Placebo: Unknown or Not Reported | 0
    Part B: Randomized - TD-9855: number analyzed (Participants) | 5
    Part B: Randomized - TD-9855: American Indian or Alaska Native | 0
    Part B: Randomized - TD-9855: Asian | 0
    Part B: Randomized - TD-9855: Native Hawaiian or Other Pacific Islander | 0
    Part B: Randomized - TD-9855: Black or African American | 0
    Part B: Randomized - TD-9855: White | 5
    Part B: Randomized - TD-9855: More than one race | 0
    Part B: Randomized - TD-9855: Unknown or Not Reported | 0
    Part C: Dose Extension: number analyzed (Participants) | 21
    Part C: Dose Extension: American Indian or Alaska Native | 0
    Part C: Dose Extension: Asian | 1
    Part C: Dose Extension: Native Hawaiian or Other Pacific Islander | 0
    Part C: Dose Extension: Black or African American | 2
    Part C: Dose Extension: White | 18
    Part C: Dose Extension: More than one race | 0
    Part C: Dose Extension: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change From Time-matched Placebo in Seated Systolic Blood Pressure (SBP)
Description: Placebo referred to the Day 1 visit, and the change from placebo referred to the time-matched difference from each TD-9855 dosing day (Days 2 through 5) relative to placebo dosing (Day 1).
Time Frame: 7 hours post-dose on Day 1 (Placebo dosing) and on each of Days 2 to 5 (TD-9855 dosing)
Population: Intent-to-treat (ITT) analysis set - All analyzable participants who received placebo on Day 1 of Part A.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Groups:
- Part A: TD-9855 1 mg: Participants who were enrolled prior to protocol amendment 2 received 1 mg of TD-9855 as an oral solution on Day 2 of the Part A treatment period.
- Part A: TD-9855 2.5 mg: Participants received 2.5 mg of TD-9855 as an oral solution on Day 2 of the Part A treatment period (Day 3 if enrolled prior to protocol amendment 2).
- Part A: TD-9855 5 mg: Participants received 5 mg of TD-9855 as an oral solution on Day 3 of the Part A treatment period (Day 4 if enrolled prior to protocol amendment 2).
- Part A: TD-9855 10 mg: Participants received 10 mg of TD-9855 as an oral solution on Day 4 of the Part A treatment period (Day 5 if enrolled prior to protocol amendment 2).
- Part A: TD-9855 20 mg: Participants received 20 mg of TD-9855 as an oral solution on Day 5 of the Part A treatment period. Participants who were enrolled prior to protocol amendment 2 were not up-titrated to the 20 mg dosing level.
Arm/Group | Part A: TD-9855 1 mg | Part A: TD-9855 2.5 mg | Part A: TD-9855 5 mg | Part A: TD-9855 10 mg | Part A: TD-9855 20 mg
Number analyzed (Participants) | 17 | 30 | 28 | 28 | 13
millimeter of mercury (mmHg) | 0.2 (18.58) | -1.8 (20.27) | -3.4 (16.50) | -2.9 (21.53) | -7.3 (18.86)

2. Primary Outcome: Part B: Change From Baseline in Seated SBP
Description: Baseline was defined as the pre-dose measurement on Day 1 of Part B.
Time Frame: Baseline and 7 hours post-dose on Day 1
Population: ITT analysis set - All analyzable participants who received any amount of placebo or TD-9855.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B: Randomized - Placebo | Part B: Randomized- TD-9855
Number analyzed (Participants) | 5 | 5
mmHg | 0.30 (27.655) | 9.00 (13.139)

3. Primary Outcome: Part C: Change From Baseline in Likert Scale Score at Week 4
Description: The Likert Scale is question 1 of the Orthostatic Hypotension Symptom Assessment (OHSA). The question asks participants to rate the severity of their orthostatic hypotension symptoms (dizziness, lightheadedness, feeling faint, or feeling like you might black out) on an 11-point scale from 0 to 10, with 0 indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference. A higher score indicates a worse outcome. Baseline was defined as the pre-lunch measurement on Day -1.
Time Frame: Baseline to Week 4
Population: ITT analysis set - All analyzable participants who received at least 1 dose of TD-9855.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part C: Dose Extension
Number analyzed (Participants) | 16
score on a scale | -2.4 (4.54)

4. Secondary Outcome: Part A and Part B: Change From Baseline in Likert Scale Score at 6 to 8 Hours
Description: The Likert Scale is question 1 of the Orthostatic Hypotension Symptom Assessment (OHSA). The question asks participants to rate the severity of their orthostatic hypotension symptoms (dizziness, lightheadedness, feeling faint, or feeling like you might black out) on an 11-point scale from 0 to 10, with 0 indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference. A higher score indicates a worse outcome. Baseline was defined as the pre-dose measurement on Day 1 for Part A and Part B. Data was collected a one point between 6 and 8 hours post-dose.
Time Frame: Baseline to a single time point between 6 to 8 hours post-dose
Population: ITT analysis set - All analyzable participants who received placebo on Day 1 of Part A. All analyzable participants who received any amount of placebo or TD-9855 in Part B.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part A: Placebo: Participants received a placebo matching TD-9855 on Day 1 of the Part A treatment period.
- Part B: Randomized - TD-9855: Part B of this study followed a randomized, double-blind, placebo-controlled, parallel design at the dose level of TD-9855 determined to have a pressor effect for a given participant in Part A. Participants from Part A were rolled over into Part B.
  Following the washout period after Part A, participants were randomized to receive a single dose of their previously tolerated dose of TD-9855 on Day 1 of the treatment period.
Arm/Group | Part A: Placebo | Part A: TD-9855 1 mg | Part A: TD-9855 2.5 mg | Part A: TD-9855 5 mg | Part A: TD-9855 10 mg | Part A: TD-9855 20 mg | Part B: Randomized - Placebo | Part B: Randomized - TD-9855
Number analyzed (Participants) | 33 | 16 | 29 | 27 | 27 | 13 | 5 | 5
score on a scale | -0.6 (2.46) | -0.9 (4.08) | -1.4 (3.61) | -1.3 (3.59) | -2.0 (3.66) | -2.2 (3.19) | -1.6 (3.44) | -1.8 (2.28)

5. Secondary Outcome: Part A and Part B: Change From Baseline in the Composite Orthostatic Hypotension Symptom Assessment (OHSA) Score
Description: The OHSA is made up of a 6-item symptoms assessment. All items were scored on an 11-point scale from 0 to 10, with 0 indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference. Activities that were marked as zero or "cannot be done for other reasons" at baseline were not included in the scoring. The composite OHSA score is the average of the response scores (for non-missing data) to the 6 questions of OHSA. A reduction in composite score indicates an improvement in symptoms. Baseline was defined as the pre-dose measurement on Day 1 for Part A and Part B. Data was collected a one point between 6 and 8 hours post-dose.
Time Frame: Baseline to a single time point between 6 to 8 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Placebo | Part A: TD-9855 1 mg | Part A: TD-9855 2.5 mg | Part A: TD-9855 5 mg | Part A: TD-9855 10 mg | Part A: TD-9855 20 mg | Part B: Randomized - Placebo | Part B: Randomized - TD-9855
Number analyzed (Participants) | 33 | 16 | 29 | 27 | 27 | 13 | 5 | 5
score on a scale | -0.07 (1.808) | -0.30 (2.157) | -0.64 (1.730) | -0.78 (2.232) | -1.22 (2.625) | -1.31 (2.340) | -1.0 (2.64) | -0.3 (1.74)

6. Secondary Outcome: Part A: Change From Time-matched Placebo in Standing SBP
Description: Placebo referred to the Day 1 visit, and the change from placebo referred to the time-matched difference from each TD-9855 dosing day (Days 2 through 5) relative to placebo dosing (Day 1). SBP was measured after 5 minutes of standing.
Time Frame: 4 and 7 hours post-dose on Day 1 (Placebo dosing) and on each of Days 2 to 5 (TD-9855 dosing)
Population: ITT analysis set - All analyzable participants who received placebo on Day 1 of Part A.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A: TD-9855 1 mg | Part A: TD-9855 2.5 mg | Part A: TD-9855 5 mg | Part A: TD-9855 10 mg | Part A: TD-9855 20 mg
Number analyzed (Participants) | 7 | 13 | 12 | 11 | 5
mmHg
  4 Hours Post-dose: number analyzed (Participants) | 6 | 13 | 12 | 11 | 5
  4 Hours Post-dose | -3.8 (8.80) | 8.6 (14.13) | 6.8 (15.85) | 8.5 (9.57) | 6.2 (3.77)
  7 Hours Post-dose: number analyzed (Participants) | 7 | 12 | 10 | 10 | 5
  7 Hours Post-dose | 12.0 (11.92) | 12.9 (20.40) | 8.9 (11.14) | 3.8 (5.94) | 0.4 (11.67)

7. Secondary Outcome: Part B: Change From Baseline in Standing SBP
Description: SBP was measured after 3 minutes of standing. Baseline was defined as the pre-dose measurement on Day 1 of Part B.
Time Frame: Baseline, 4 and 7 hours post-dose on Day 1
Population: ITT analysis set - All analyzable participants who received any amount of placebo or TD-9855.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B: Randomized - Placebo | Part B: Randomized- TD-9855
Number analyzed (Participants) | 3 | 2
mmHg
  4 Hours Post-dose: number analyzed (Participants) | 2 | 2
  4 Hours Post-dose | -5.0 (8.49) | 20.5 (2.12)
  7 Hours Post-dose | -4.0 (12.00) | 21.5 (9.19)

8. Secondary Outcome: Part A: Change From Time-matched Placebo in Seated SBP
Description: as for outcome 1
Time Frame: 4, 7, 9, 12 hours post-dose on Day 1 (placebo) and Days 2 to 5 (TD-9855 dosing)
Population: ITT analysis set - All analyzable participants who received placebo on Day 1 of Part A.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A: TD-9855 1 mg | Part A: TD-9855 2.5 mg | Part A: TD-9855 5 mg | Part A: TD-9855 10 mg | Part A: TD-9855 20 mg
Number analyzed (Participants) | 17 | 31 | 28 | 28 | 13
mmHg
  4 Hours Post-dose | -3.2 (15.89) | 2.4 (15.24) | 5.9 (21.85) | 4.9 (20.14) | 0.7 (17.40)
  7 Hours Post-dose: number analyzed (Participants) | 17 | 30 | 28 | 28 | 13
  7 Hours Post-dose | 0.2 (18.58) | -1.8 (20.27) | -3.4 (16.50) | -2.9 (21.53) | -7.3 (18.86)
  9 Hours Post-dose: number analyzed (Participants) | 17 | 29 | 28 | 28 | 13
  9 Hours Post-dose | 4.1 (19.08) | 0.7 (18.90) | 5.5 (21.14) | 2.5 (20.85) | 9.8 (26.48)
  12 Hours Post-dose: number analyzed (Participants) | 16 | 28 | 27 | 27 | 13
  12 Hours Post-dose | 2.4 (22.20) | -1.4 (17.44) | 0.4 (19.86) | 7.4 (24.88) | -2.5 (14.42)

9. Secondary Outcome: Part B: Change From Baseline in Seated SBP
Description: Baseline was defined as the pre-dose measurement on Day 1 of Part B.
Time Frame: Baseline and 4, 7, 9 and 12 hours post-dose on Day 1
Population: ITT analysis set - All analyzable participants who received any amount of placebo or TD-9855.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part B: Randomized - Placebo | Part B: Randomized- TD-9855
Number analyzed (Participants) | 5 | 5
mmHg
  4 Hours Post-dose | -9.70 (26.397) | 11.20 (26.407)
  7 Hours Post-dose | 0.30 (27.665) | 9.00 (13.139)
  9 Hours Post-dose | 6.70 (29.668) | 7.40 (19.415)
  12 Hours Post-dose | 9.90 (32.809) | -6.90 (43.118)

10. Secondary Outcome: Part A: Change From Time-matched Placebo in Duration of Standing During the Orthostatic Standing Test (OST)
Description: Blood pressure (BP) and heart rate (HR) measurements were recorded with automated (or manual) sphygmomanometer, after being seated for 5 min and 10 min, and after standing for 1, 3, 5, and 10 min. The standing time was measured with a chronometer and the duration of standing was recorded. The total duration of standing may have occurred between 2 of the predefined time points, or the participant may have been able to stand for longer than the 10-min standing test. In either case, the total duration was recorded. Placebo referred to the Day 1 visit, and the change from placebo referred to the time-matched difference from each TD-9855 dosing day (Days 2 through 5) relative to placebo dosing (Day 1) of Part A.
Time Frame: 4 and 7 hours post-dose on Day 1 (Placebo dosing) and on each of Days 2 to 5 (TD-9855 dosing)
Population: ITT analysis set - All analyzable participants who received placebo on Day 1 of Part A.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part A: TD-9855 1 mg | Part A: TD-9855 2.5 mg | Part A: TD-9855 5 mg | Part A: TD-9855 10 mg | Part A: TD-9855 20 mg
Number analyzed (Participants) | 17 | 31 | 28 | 28 | 13
minutes
  4 Hours Post-dose | 0.698 (3.1357) | 0.799 (2.7898) | 1.085 (3.4188) | 1.579 (3.5527) | 1.081 (2.8553)
  7 Hours Post-dose: number analyzed (Participants) | 16 | 29 | 27 | 27 | 13
  7 Hours Post-dose | 0.747 (3.3856) | 1.343 (2.7847) | 0.952 (3.6232) | 0.986 (4.3645) | 1.159 (2.8264)

11. Secondary Outcome: Part B: Change From Baseline in Duration of Standing During the OST
Description: BP and heart rate HR measurements were recorded with automated (or manual) sphygmomanometer, after being seated for 5 min and 10 min, and after standing for 1, 3, 5, and 10 min. The standing time was measured with a chronometer and the duration of standing was recorded. The total duration of standing may have occurred between 2 of the predefined time points, or the participant may have been able to stand for longer than the 10-min standing test. In either case, the total duration was recorded. Baseline was defined as the predose measurement on Day 1 of Part B.
Time Frame: Baseline and 7 hours post-dose on Day 1
Population: ITT analysis set - All analyzable participants who received any amount of placebo or TD-9855.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part B: Randomized - Placebo | Part B: Randomized- TD-9855
Number analyzed (Participants) | 5 | 5
minutes | 3.38 (5.275) | 0.15 (0.5080)
Statistical Analysis 1: Comparison: Part B: Randomized - Placebo vs Part B: Randomized- TD-9855; Least squares mean differences were calculated based on a repeated-measures mixed-effect model with change from baseline at different time points as the dependent variable, the treatment group (TD-9855 or placebo), time point, baseline and the interaction between the treatment group and time point as fixed factors. A compound symmetry was used as the variance-covariance structure; Test type: Superiority; p = 0.0399, Repeated-measures Mixed-effect Model — P-values were reported without multiplicity adjustment; Least Squares Mean Difference = -4.40, 95% CI 2-sided [-8.57 to -0.23]

12. Secondary Outcome: Part C: Change From Baseline in the Composite OHSA Score
Description: The OHSA is made up of a 6-item symptoms assessment. All items were scored on an 11-point scale from 0 to 10, with 0 indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference, and the option of selecting "cannot be done for other reasons." Activities that were marked as zero or "cannot be done for other reasons" at baseline were not included in the scoring. The composite OHSA score is the average of the response scores (for non-missing data) to the 6 questions of OHSA. Baseline was defined as the pre-lunch measurement on Day -1.
Time Frame: Baseline to Day 169
Population: ITT analysis set - All analyzable participants who received at least 1 dose of TD-9855.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part C: Dose Extension
Number analyzed (Participants) | 16
score on a scale
  Day 29 | -0.97 (2.780)
  Day 57 | -0.78 (2.726)
  Day 85: number analyzed (Participants) | 13
  Day 85 | -0.45 (2.276)
  Day 113: number analyzed (Participants) | 13
  Day 113 | -1.33 (2.556)
  Day 140: number analyzed (Participants) | 11
  Day 140 | -1.36 (2.537)
  Day 155: number analyzed (Participants) | 11
  Day 155 | -0.21 (3.203)
  Day 169: number analyzed (Participants) | 10
  Day 169 | 0.55 (2.467)

13. Secondary Outcome: Part C: Change From Baseline in the Orthostatic Hypotension Daily Activity Scale (OHDAS)
Description: The OHDAS is made up of a 4-item daily activity assessment. All items were scored on an 11-point scale from 0 to 10, with 0 indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference, and the option of selecting "cannot be done for other reasons." Activities that were marked as zero or "cannot be done for other reasons" at baseline were not included in the scoring. The composite OHDAS score is the average of the response scores (for non-missing data) to the 4 questions of OHDAS. Baseline was defined as the pre-lunch measurement on Day -1.
Time Frame: Baseline to Day 169
Population: ITT analysis set - All analyzable participants who received at least 1 dose of TD-9855.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part C: Dose Extension
Number analyzed (Participants) | 16
score on a scale
  Day 29 | -1.12 (2.889)
  Day 57 | -1.49 (2.438)
  Day 85: number analyzed (Participants) | 13
  Day 85 | -2.11 (2.398)
  Day 113: number analyzed (Participants) | 13
  Day 113 | -1.63 (2.424)
  Day 140: number analyzed (Participants) | 11
  Day 140 | -1.83 (2.610)
  Day 155: number analyzed (Participants) | 11
  Day 155 | -0.86 (3.328)
  Day 169: number analyzed (Participants) | 10
  Day 169 | -0.69 (2.509)

14. Secondary Outcome: Part C: Change From Baseline in the Orthostatic Hypotension Questionnaire (OHQ) Score
Description: The OHQ is a 2-component questionnaire made up of 6-item symptoms assessment referred to as OHSA, and a 4-item daily activity assessment referred to as the OHDAS. All items were scored on an 11-point scale from 0 to 10, with 0 indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference, and the option of selecting "cannot be done for other reasons." Activities that were marked as zero or "cannot be done for other reasons" at baseline were not included in the scoring.
  The composite OHSA score is the average of the response scores (for non-missing data) to the 6 questions of OHSA. The composite OHDAS score is the average of the response scores (for non-missing data) to the 4 questions of OHDAS. The OHQ composite score is the average of the OHSA and OHDAS composite scores.
  Baseline was defined as the pre-lunch measurement on Day -1.
Time Frame: Baseline to Day 169
Population: ITT analysis set - All analyzable participants who received at least 1 dose of TD-9855.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part C: Dose Extension
Number analyzed (Participants) | 16
score on a scale
  Day 29 | -1.04 (2.531)
  Day 57 | -1.14 (2.290)
  Day 85: number analyzed (Participants) | 13
  Day 85 | -1.28 (1.966)
  Day 113: number analyzed (Participants) | 13
  Day 113 | -1.48 (2.253)
  Day 140: number analyzed (Participants) | 11
  Day 140 | -1.60 (2.273)
  Day 155: number analyzed (Participants) | 11
  Day 155 | -0.53 (3.0711)
  Day 169: number analyzed (Participants) | 10
  Day 169 | -0.07 (2.276)

15. Secondary Outcome: Part C: Change From Baseline in Standing SBP
Description: SBP was measured after 3 minutes of standing. Baseline was defined as the pre-lunch measurement on Day 1.
Time Frame: Baseline to Day 169
Population: ITT analysis set - All analyzable participants who received at least 1 dose of TD-9855.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part C: Dose Extension
Number analyzed (Participants) | 11
mmHg
  Day 1 | 15.5 (14.711)
  Day 29: number analyzed (Participants) | 10
  Day 29 | 7.6 (22.37)
  Day 85: number analyzed (Participants) | 9
  Day 85 | 23.0 (19.21)
  Day 140: number analyzed (Participants) | 7
  Day 140 | 21.0 (44.03)
  Day 155: number analyzed (Participants) | 6
  Day 155 | 23.2 (43.64)
  Day 169: number analyzed (Participants) | 5
  Day 169 | 47.2 (52.18)

16. Secondary Outcome: Part C: Change From Baseline in Seated SBP
Description: Baseline was defined as the pre-breakfast measurement on Day 1.
Time Frame: Baseline to Day 169
Population: ITT analysis set - All analyzable participants who received at least 1 dose of TD-9855.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part C: Dose Extension
Number analyzed (Participants) | 21
mmHg
  Day 1 | 11.19 (23.792)
  Day 29: number analyzed (Participants) | 16
  Day 29 | 7.56 (26.487)
  Day 85: number analyzed (Participants) | 13
  Day 85 | 7.81 (25.109)
  Day 140: number analyzed (Participants) | 11
  Day 140 | 13.36 (33.787)
  Day 155: number analyzed (Participants) | 11
  Day 155 | 15.23 (23.648)
  Day 169: number analyzed (Participants) | 10
  Day 169 | 12.10 (35.624)

17. Secondary Outcome: Part C: Change From Baseline in Duration of Standing During the OST
Description: BP and heart rate HR measurements were recorded with automated (or manual) sphygmomanometer, after being seated for 5 min and 10 min, and after standing for 1, 3, 5, and 10 min. The standing time was measured with a chronometer and the duration of standing was recorded. The total duration of standing may have occurred between 2 of the predefined time points, or the participant may have been able to stand for longer than the 10-min standing test. In either case, the total duration was recorded. Baseline was defined as the pre-breakfast measurement on Day 1.
Time Frame: Baseline to Day 169
Population: ITT analysis set - All analyzable participants who received at least 1 dose of TD-9855.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part C: Dose Extension
Number analyzed (Participants) | 21
minutes
  Day 1 | 0.942 (4.2861)
  Day 29: number analyzed (Participants) | 16
  Day 29 | 1.328 (3.4217)
  Day 85: number analyzed (Participants) | 13
  Day 85 | 4.069 (6.6833)
  Day 140: number analyzed (Participants) | 11
  Day 140 | 4.380 (6.1494)
  Day 155: number analyzed (Participants) | 11
  Day 155 | 4.533 (7.3741)
  Day 169: number analyzed (Participants) | 10
  Day 169 | 1.923 (7.3697)

18. Secondary Outcome: Part C: Change From Baseline in Supine SBP to Seated SBP
Description: Baseline is defined as pre-breakfast measurement on Day 1. The difference in SBP from a supine to a seated position was measured at baseline and at each time point. The change from baseline was calculated at each time point.
Time Frame: Baseline to Day 169
Population: ITT analysis set - All analyzable participants who received at least 1 dose of TD-9855.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part C: Dose Extension
Number analyzed (Participants) | 21
mmHg
  Day 1 Pre-lunch | 5.60 (13.245)
  Day 2 Pre-breakfast | -2.60 (20.689)
  Day 2 Pre-lunch | 2.76 (12.802)
  Day 15 Pre-breakfast: number analyzed (Participants) | 17
  Day 15 Pre-breakfast | 5.09 (17.448)
  Day 15 Pre-lunch: number analyzed (Participants) | 17
  Day 15 Pre-lunch | 10.03 (14.842)
  Day 29 Pre-breakfast: number analyzed (Participants) | 16
  Day 29 Pre-breakfast | 9.38 (17.736)
  Day 29 Pre-lunch: number analyzed (Participants) | 16
  Day 29 Pre-lunch | 3.53 (15.174)
  Day 85 Pre-breakfast: number analyzed (Participants) | 13
  Day 85 Pre-breakfast | 2.19 (15.788)
  Day 85 Pre-lunch: number analyzed (Participants) | 13
  Day 85 Pre-lunch | 4.38 (21.349)
  Day 140 Pre-breakfast: number analyzed (Participants) | 11
  Day 140 Pre-breakfast | 0.73 (19.159)
  Day 140 Pre-lunch: number analyzed (Participants) | 11
  Day 140 Pre-lunch | 1.82 (18.000)
  Day 155 Pre-breakfast: number analyzed (Participants) | 11
  Day 155 Pre-breakfast | 2.68 (23.703)
  Day 155 Pre-lunch: number analyzed (Participants) | 11
  Day 155 Pre-lunch | 1.36 (19.694)
  Day 169 Pre-breakfast: number analyzed (Participants) | 10
  Day 169 Pre-breakfast | 1.50 (14.650)
  Day 169 Pre-lunch: number analyzed (Participants) | 10
  Day 169 Pre-lunch | 2.95 (18.669)

ADVERSE EVENTS:
Time Frame: Part A: Day 1 to Day 6 of Part A treatment period, plus 30 days. Part B: Day 1 of Part B treatment period, plus 30 days. Part C: Day 1 to Day 169 of Part C treatment period.
Arm/Group | Part A: Placebo | Part A: TD-9855 1 mg | Part A: TD-9855 2.5 mg | Part A: TD-9855 5 mg | Part A: TD-9855 10 mg | Part A: TD-9855 20 mg | Part B: Randomized - Placebo | Part B: Randomized - TD-9855 | Part C: Dose Extension
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/17 | 0/31 | 0/29 | 0/28 | 0/13 | 0/5 | 0/5 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/17 | 0/31 | 0/29 | 0/28 | 0/13 | 0/5 | 0/5 | 5/21
Other Adverse Events (participants affected / at risk) | 7/34 | 4/17 | 5/31 | 3/29 | 6/28 | 1/13 | 0/5 | 1/5 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=34) | Part A: TD-9855 1 mg (N=17) | Part A: TD-9855 2.5 mg (N=31) | Part A: TD-9855 5 mg (N=29) | Part A: TD-9855 10 mg (N=28) | Part A: TD-9855 20 mg (N=13) | Part B: Randomized - Placebo (N=5) | Part B: Randomized - TD-9855 (N=5) | Part C: Dose Extension (N=21)
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=34) | Part A: TD-9855 1 mg (N=17) | Part A: TD-9855 2.5 mg (N=31) | Part A: TD-9855 5 mg (N=29) | Part A: TD-9855 10 mg (N=28) | Part A: TD-9855 20 mg (N=13) | Part B: Randomized - Placebo (N=5) | Part B: Randomized - TD-9855 (N=5) | Part C: Dose Extension (N=21)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 3
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impulse-control disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised infection (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ear canal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Part B of the study was discontinued in protocol amendment 2, however details regarding Part B are still included in this summary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT02705755/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT02705755/SAP_001.pdf